CLINICAL TRIAL: NCT06566794
Title: KF2022#4-tutkimus:Beetasalpaajan ja tulehduskipulääkkeen Vaikutus CYP-entsyymivälitteiseen lääkeainemetaboliaan
Brief Title: KF2022#4-trial: Effects of a Beta Blocker and NSAID on CYP Mediated Drug Metabolism
Acronym: KF2022#4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Janne Backman, Professor, Head physician, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KF2022#4; 2023-000002-25 (EudraCT Number)
Record Dates: First submitted 2024-08-04; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Caffeine; Bupropion; Capsules; repaglinide; Flurbiprofen; Omeprazole; Dextromethorphan; Solutions; Midazolam; Simvastatin; Tablets; Carvedilol; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo tablets (2 x Placebo) and 150 ml water at 8.00 a.m. on the study day.
  Study drug doses (caffeine 50 mg, bupropion 20 mg, repaglinide 0,05 mg, flurbiprofen 10 mg, omeprazole 10 mg, dextromethorphan 10 mg, midazolam 1,0 mg, simvastatin 10 mg) and 250 ml water at 9:00 a.m.
  Interventions: Drug: Caffeine Tablet; Drug: Bupropion Hydrochloride Capsels; Drug: Repaglinide Capsels; Drug: Flurbiprofen Capsels; Drug: Omeprazole 10 MG; Drug: Dextromethorphan Oral Solution; Drug: Midazolam oral solution; Drug: Simvastatin tablets; Drug: Placebo
- Carvedilol (Active Comparator): Carvedilol tablets (2 x Carvedilol STADA 25 mg) and 150 ml water at 8.00 a.m. on the study day.
  Study drug doses (caffeine 50 mg, bupropion 20 mg, repaglinide 0,05 mg, flurbiprofen 10 mg, omeprazole 10 mg, dextromethorphan 10 mg, midazolam 1,0 mg, simvastatin 10 mg) and 250 ml water at 9:00 a.m.
  Interventions: Drug: Caffeine Tablet; Drug: Bupropion Hydrochloride Capsels; Drug: Repaglinide Capsels; Drug: Flurbiprofen Capsels; Drug: Omeprazole 10 MG; Drug: Dextromethorphan Oral Solution; Drug: Midazolam oral solution; Drug: Simvastatin tablets; Drug: Carvedilol
- Diclofenac (Active Comparator): Diclofenac tablet (1 x Voltaren Rapid 50 mg) three times a day around 8.00 a.m., 3.00 p.m. and 9.00 p.m. for three days.
  Diclofenac tablet (1 x Voltaren Rapid 50 mg) and 150 ml water at 8.00 a.m., 3.00 p.m. and 9.00 p.m. on the study day (3rd day of diclofenac treatment).
  Study drug doses (caffeine 50 mg, bupropion 20 mg, repaglinide 0,05 mg, flurbiprofen 10 mg, omeprazole 10 mg, dextromethorphan 10 mg, midazolam 1,0 mg, simvastatin 10 mg) and 250 ml water at 9:00 a.m.
  Interventions: Drug: Caffeine Tablet; Drug: Bupropion Hydrochloride Capsels; Drug: Repaglinide Capsels; Drug: Flurbiprofen Capsels; Drug: Omeprazole 10 MG; Drug: Dextromethorphan Oral Solution; Drug: Midazolam oral solution; Drug: Simvastatin tablets; Drug: Diclofenac

INTERVENTIONS:
Drug: Caffeine Tablet — 0,5 x 100 mg tablet (50 mg caffeine).
  Other Names: YA Kofeiinitabletti 100 mg, Yliopiston apteekki
Drug: Bupropion Hydrochloride Capsels — 1 x 20 mg tablet.
  Other Names: Bupropion hydrochloride 20 mg caps, HUS Apteekki
Drug: Repaglinide Capsels — 1 x 0,05 mg tablet.
  Other Names: Repaglinide 0.05 mg caps, HUS Apteekki
Drug: Flurbiprofen Capsels — 1 x 10 mg tablet.
  Other Names: Flurbiprofen 10 mg caps, HUS Apteekki
Drug: Omeprazole 10 MG — 1 x 10 mg tablet.
  Other Names: Losec Mups 10 mg enterotablet, AstraZeneca
Drug: Dextromethorphan Oral Solution — 5,0 ml of 2 mg/ml oral solution (10 mg dextromethorphan).
  Other Names: Rometor Ratiopharm 2 mg/ml oral solution, Ratiopharm
Drug: Midazolam oral solution — 0,5 ml of 2 mg/ml oral solution (1,0 mg midazolam).
  Other Names: Midazolam-Ratiopharm 2 mg/ml oral solution, Ratiopharm
Drug: Simvastatin tablets — 1 x 10 mg tablet.
  Other Names: Simvastatin Krka 10 mg tablet, KRKA
Drug: Placebo — 2 x placebo tablets in the Placebo Phase/Arm
  Other Names: Placebo, 9 mm tablet, Yliopiston apteekki
  Arms: Placebo
Drug: Carvedilol — 2 x 25 mg tablets
  Other Names: Carvedilol STADA 25 mg tablet, STADA Arzneimittel AG
  Arms: Carvedilol
Drug: Diclofenac — 1 x 50 mg tablet (three times daily for three days)
  Other Names: Voltaren Rapid 50 mg, Novartis Finland Oy
  Arms: Diclofenac

SUMMARY:
Carvedilol is a non-selective beta-blocker in common clinical use, used to treat hypertension, heart failure, and angina pectoris symptoms associated with coronary artery disease. Diclofenac is a non-selective anti-inflammatory drug in general use, which is used to treat rheumatic diseases, osteoarthritis, musculoskeletal pain conditions, menstrual pains and migraines, among others. In our recent experiments involving liver cell enzymes, both carvedilol and diclofenac were found to inhibit several cytochrome P450 (CYP) enzymes central to drug metabolism, potentially leading to adverse drug interactions with other drugs metabolized by the same enzyme. The purpose of this study is to investigate the effects of the use of carvedilol and diclofenac on the activity of key CYP enzymes in drug metabolism in healthy volunteers using a low-dose model drug combination covering seven CYP enzymes.

In an open three-phase, randomized, crossover study with 12 healthy volunteers, the subjects will receive a drug combination of caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam and simvastatin and as a premedication either placebo, carvedilol or diclofenac. Blood samples will be collected and carvedilol, diclofenac, caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam and simvastatin pharmacokinetics will be monitored up to 23 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-40
* Healthy
* Systolic blood pressure ≥110 mmHg
* Heart rate ≥ 55/min
* Normal ECG
* Accepted results from laboratory tests (blood haemoglobin, basic blood count and blood platelets, alanine aminotransferase, alkaline phosphatase, glutamyl transferase, creatine kinase, creatinine, plasma glucose concentration, plasma potassium and sodium). Negative pregnancy test result (serum human chorionic gonadotropin) for women.

Exclusion Criteria:

* Significant disease
* Previous or current gastrointestinal bleeding, ulcer or perforation
* Findings of a medical examination and laboratory tests, which require a more detailed examination of the state of health
* Smoking
* Hormonal birth control or other regular medication
* Pregnancy (current or planned) or nursing
* Participation in any other studies involving investigational or marketed drug products within three months prior to the entry into this study
* Donation of blood within three months prior to the entry into this study
* Significant overweight / small or hard-to-find veins
* BMI < 18.5 kg/m2
* Insufficient Finnish language skills
* Hypersensitivity or contraindication to study drugs

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration - time curve of carvedilol, diclofenac, caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam and simvastatin | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 23 hours after administration the drugs.

SECONDARY OUTCOMES:
Peak plasma concentration for carvedilol, diclofenac, caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam, simvastatin and their metabolites. | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 23 hours after administration the drugs.
Half-life for carvedilol, diclofenac, caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam, simvastatin and their metabolites. | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 23 hours after administration the drugs.
Time to peak plasma concentration for carvedilol, diclofenac, caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam, simvastatin and their metabolites. | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 23 hours after administration the drugs.
Fractional areas under concentration-time curve (AUC) for carvedilol, diclofenac, caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam, simvastatin and their metabolites. | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 23 hours after administration the drugs.
Areas under concentration-time curve (AUC) for carvedilol, diclofenac, caffeine, bupropion, repaglinide, flurbiprofen, omeprazole, dextromethorphan, midazolam, simvastatin and their metabolites. | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 23 hours after administration the drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No